CLINICAL TRIAL: NCT01156298
Title: Phase IV, Multi-center, Non-treatment, Observational, Registry Study to Determine Long Term Effects of AVONEX® Therapy on EDSS, MRI, QoL, and Cognition.
Brief Title: Controlled High Risk AVONEX® Multiple Sclerosis Prevention Study In Ongoing Neurological Surveillance
Acronym: CHAMPIONS CONT
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Biogen (Industry)
Responsible Party: Project Manager, Biogen Idec Inc.
Other Study IDs: 004-09-AVX
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Patients were diagnosed upon entry into CHAMPS with CIS demyelinating event with MRI lesions consistent with MS. Patients are eligible regardless of whether they have converted to Clinically Definite Multiple Sclerosis (CDMS) or not. Cohort 1 patients will have annual EDSS, self-report EDSS, medication review and relapse recalculation. SF-36 and SDMT assessments will be performed at years 1 and 5 during routine office visits. A MRI will be performed each patient's 15 year anniversary date.
- Cohort 2: Patients were diagnosed upon entry into CHAMPS with CIS demyelinating event with MRI lesions consistent with MS. Patients are eligible regardless of whether they have converted to Clinically Definite Multiple Sclerosis (CDMS) or not. Patients will be waiving written informed consent and asked to provide concomitant medication, self-reported EDSS, and SF-36 only.

SUMMARY:
Phase IV, multi-center, non-treatment, observational, registry study to determine long term effects of AVONEX® therapy on EDSS, MRI, QoL, and cognition.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the impact of long term AVONEX® treatment on physical status, measured by expanded disability scale score (EDSS), of patients with Multiple Sclerosis (MS) after their first clinical event (clinically isolated syndrome) and Magnetic Resonance Imaging (MRI) consistent with MS.

Secondary objectives are to determine the impact of long term therapy with AVONEX® on the following:

a) MRI parameters- new or enlarging T2 lesions, T2 lesion volume, T1 lesion volume, brain parenchymal fraction (BPF) b) Quality of Life (QoL): Heath Status Questionnaire (SF-36) c) Symbol Digit Modality Test (SDMT)

2. To determine the long term impact of therapy on the following in patients treated at the onset of clinically isolated event (CIS)

1. EDSS
2. MRI parameters
3. SF-36
4. SDMT

   3. To determine early clinical and MRI predictors of disease progression.

   Approximately 383 patients participated in CHAMPS, the original AVONEX® placebo trial, will be approached for study participation. The patient population will be divided into two cohorts.

   Cohort 1: Patients that participated in CHAMPS and CHAMPIONS 10 will be approached for study participation at approximately twenty-four CHAMPIONS Continuation investigative sites.

   Cohort 2: Patients that participated in CHAMPS will be located and approached for study participation. Patient that participated in CHAMPIONS 10 will not be excluded from Cohort 2. Efforts will be made to potentially locate patients through either the original CHAMPS investigative sites, through the Biogen Idec patient services database, and/or a third party (i.e., patient location service vendor) or some combination of the three. .

   For both cohorts, public databases may be utilized for patient reported death.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be screened for this study if all of the following criteria are met:

  1. All patients must have been originally enrolled in CHAMPS, regardless of randomization arm. Only Cohort 1 patients must have been enrolled in CHAMPIONS 10.
  2. Willing and able to provide informed consent (Cohort 1), waiver of informed consent (Cohort 2), or reported patient death through public database search.
  3. Ability to read and write English (patient reported assessment tools are in English only).

Exclusion Criteria:

* Candidates will be excluded from study screening if any of the following exclusion criteria exist:

  1. Patients not participating in the original CHAMPS study.
  2. Alternative diagnosis to MS discovered.
  3. Patient unwilling or unable to provide informed consent (Cohort 1) or waiver of informed consent (Cohort 2), as applicable.
  4. Any other reasons that, in the opinion of the Investigator (Cohort 1) or Patient Coordination Center (Cohort 2), the patient is determined to be unsuitable for enrollment into this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 383 patients participated in CHAMPS, the original AVONEX® placebo trial, will be approached for study participation. The patient population will be divided into two cohorts.
  Cohort 1: Patients that participated in CHAMPS and CHAMPIONS 10 will be approached for study participation at approximately twenty-four CHAMPIONS Continuation investigative sites. Patients were diagnosed upon entry into CHAMPS with CIS demyelinating event with MRI lesions consistent with MS. Patients are eligible regardless of whether they have converted to Clinically Definite Multiple Sclerosis (CDMS) or not. Cohort 1 patients will have annual EDSS, self-report EDSS, medication review and relapse recalculation. SF-36 and SDMT assessments will be performed at years 1 and 5 during routine office visits. A MRI will be performed each patient's 15 year anniversary date. See Schedule of Assessments, section 12.
  Cohort 2: Patients that participated in CHAMPS will be located and approached for s
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
EDSS | yearly
MRI | last visit, 15 year anniversary

SECONDARY OUTCOMES:
Quality of Life | year 1 & 5
Symbol Digit Modality Test | year 1 & 5

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Buffalo, New York, United States